CLINICAL TRIAL: NCT02636426
Title: Sorafenib Administered Using a High-dose, Pulsatile Regimen in Patients With Advanced Solid Malignancies: a Phase I Exposure Escalation Study
Brief Title: Sorafenib Administered Using a High-dose, Pulsatile Regimen: a Phase I Exposure Escalation Study
Acronym: SOPRANO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, H.M.W. Verheul, Prof. Dr. MD PhD, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015.224
Record Dates: First submitted 2015-12-02; First posted 2015-12-21 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms
Keywords: phase I study; sorafenib; high-dose schedule; pharmacokinetics; drug monitoring
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib (Experimental): In this phase I study patients are treated with high-dose, pulsatile sorafenib in escalating AUC0-12h cohorts.
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — In new dosing schedule of sorafenib is investigated in this study: high-dose, pulsatile sorafenib
  Other Names: Nexavar

SUMMARY:
Sorafenib is an oral anticancer drug and inhibits multiple protein kinases important for tumor growth and metastases, including VEGFR, PDGFR, and RAF kinases. In daily clinical practice it is currently used at a dose of 400 mg twice daily in a continuous schedule. In this phase I study patients will be treated with a new dosing schedule of sorafenib: i.e. a high-dose, pulsatile schedule. The tolerability and safety of this new schedule is examined in exposure escalation cohorts based on a target plasma AUC0-12h (area under the curve). Exposure escalation cohorts are used instead of conventional dose escalation cohorts because the effect of a drug is dependent of its AUC levels and large differences in plasma sorafenib AUC0-12h have previously been shown between patients treated at the same dose level. Using pharmacokinetic monitoring, the sorafenib dose will be adjusted to a target plasma AUC0-12h. The escalation cohorts consist of 3-6 patients per exposure level starting with a target plasma sorafenib AUC0-12h level of 25-50 mg/L/h. After the determination of the maximum tolerated AUC0-12h, 10 additional patients will be entered into an expansion cohort. In the expansion cohort the patients will be treated with a weekly pulse of sorafenib at the maximum tolerated AUC0-12h for further assessment of safety and preliminary exploration of efficacy.

DETAILED DESCRIPTION:
Rationale: Preclinical research showed improved efficacy of sorafenib when given in a high-dose, pulsatile schedule compared with conventional (lower dose) continuous scheduling as a result of higher peak concentrations in the tumor. In this phase I study patients will be treated with high-dose, pulsatile sorafenib in exposure escalation cohorts. Exposure escalations cohorts are based on a target plasma AUC0-12h (area under the curve) and are used instead of conventional dose escalation cohorts because the effect of a drug is dependent of its AUC levels and large differences in plasma sorafenib AUC0-12h have previously been shown between patients treated at the same dose level.

Primary Objectives:

* To determine the maximum tolerated plasma AUC0-12h of high-dose sorafenib administered in a weekly, pulsatile schedule.
* To assess the safety and tolerability of high-dose, pulsatile sorafenib.

Secondary Objectives:

* To determine the pharmacokinetic behaviour of sorafenib and its major active metabolite pyridine N-oxide when administered in a weekly, pulsatile schedule.
* To determine a recommended phase II plasma AUC0-12h of high-dose sorafenib in a weekly pulsatile schedule.
* Preliminary assessment of the efficacy of high-dose, pulsatile sorafenib administered at the maximum tolerated plasma AUC0-12h.
* To determine skin and intratumoral concentrations of sorafenib and their correlation with plasma and whole blood concentrations.
* To select 1-2 optimal time points from the AUC0-12h data to determine sorafenib exposure using a finger puncture.

Study design: A single center, open-label, phase I study of high-dose, pulsatile sorafenib administered in exposure escalation cohorts.

Study population: Adult patients with locally advanced or metastatic disease for whom no standard therapy exists.

Treatment: Patients will be treated in exposure escalation cohorts with high-dose sorafenib administered in a weekly pulsatile schedule. Using pharmacokinetic monitoring, the sorafenib dose will be adjusted to a target plasma AUC0-12h. The escalation cohorts consist of 3-6 patients per exposure level starting with a target plasma sorafenib AUC0-12h level of 25-50 mg/L/h. After the determination of the maximum tolerated AUC0-12h, 10 additional patients will be entered into an expansion cohort. In the expansion cohort the patients will be treated with a weekly pulse of sorafenib at the maximum tolerated AUC0-12h for further assessment of safety and preliminary exploration of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological documentation of incurable locally advanced or metastatic solid malignancy for which no standard therapy exists.
2. Patients eligible for the expansion cohort must be willing to undergo tumor and skin biopsies, while tumor and skin biopsies are optional for patients enrolled in the escalation cohort. Primary tumor or metastatic site must be accessible for biopsy. Bone metastases are excluded as a biopsy site.
3. Evaluable disease by RECIST version 1.1. criteria (see appendix III; at least 1 target or non-target lesion for the dose escalation cohorts; at least 1 target lesion the for dose expansion cohorts).
4. Patients must have documented radiographic or clinical progressive disease.
5. Age ≥ 18 years.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 (appendix IV).
7. Normal 12-lead ECG (clinically insignificant abnormalities permitted), and left ventricular ejection fraction (LVEF) > 50% evaluated by multigated acquisition scan (MUGA) or echocardiogram.
8. Normal or regulated thyroid function - supplementation or blocking drugs permitted.
9. Urine analysis: no clinically significant abnormalities.
10. Albumin higher than 25 g/L.
11. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 14 days prior to screening:

    * Hemoglobin ≥ 5,6 mmol/L
    * Absolute neutrophil count (ANC) ≥ 1,5 x 10*9/l
    * Platelet count ≥ 100 x 10*9/l
    * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). Patients with known Gilbert's disease who have serum bilirubin ≤ 3x ULN may be enrolled.
    * ALT and AST ≤ 2.5 x ULN (in case of liver metastases: ≤ 5 times ULN).
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (based on MDRD).
    * PT-INR/PTT < 1.5 x ULN, unless coumarin derivatives are used.
    * Activated partial thromboplastin time < 1.25 x ULN (therapeutic anticoagulation therapy is allowed, if this treatment can be interrupted for a biopsy as judged by the treating physician).

Exclusion Criteria:

1. Evidence of a significant uncontrolled concomitant disease, such as cardiovascular disease (including stroke, New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to screening, unstable arrhythmia, clinically significant valvular heart disease and unstable angina); nervous system, pulmonary (including obstructive pulmonary disease and history of symptomatic bronchospasm), renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture.
2. Prior radiotherapy in the abdominal or thoracic area or in > 3 vertebrae in the spine (if long interval since previous radiotherapy or radiotherapy in ≤ 3 vertebrae, eligibility will be decided on an individual basis by the primary investigator).
3. Poorly controlled hypertension despite adequate blood pressure medication. Blood pressure must be ≤ 160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 2 separate measurements.
4. Seizure disorders requiring anticonvulsant therapy.
5. Major surgery, other than diagnostic surgery, within 4 weeks prior to day 1, without complete recovery.
6. Known active bacterial, viral, fungal, mycobacterial, or other infection (including HIV and atypical mycobacterial disease, but excluding fungal infection of the nail beds).
7. Known hypersensitivity to sorafenib or to its excipients.
8. Presence of any significant central nervous system or psychiatric disorder(s) that would interfere with the patient's compliance.
9. Drug or alcohol abuse.
10. Any evidence of a disease or condition that might affect compliance with the protocol or interpretation of the study results or render the patient at high risk from treatment complications.
11. Unwillingness or inability to comply with study and follow-up procedures.
12. Chemotherapy, radiotherapy, or biologic therapy within the previous 4 weeks; Nitrosoureas or mitomycin C within the previous 6 weeks; Investigational agents within the previous 4 weeks.
13. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.
14. Untreated or active central nervous system (CNS) metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control).
15. Patients with a history of treated CNS metastases are eligible, provided that all of the following criteria are met:

    * Presence of evaluable or measurable disease outside the CNS
    * Radiographic demonstration of stabilization upon completion of CNS-directed therapy and no evidence of interim progression between completion of CNS-directed therapy and the screening radiographic study
    * Completion of radiotherapy ≥ 8 weeks prior to the screening radiographic study
    * Discontinuation of corticosteroids and anticonvulsants ≥ 4 weeks prior to the screening radiographic study
16. Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative pregnancy test performed within 7 days of the start of treatment. Both men and women enrolled in this trial must agree to use adequate barrier birth control measures (e.g., cervical cap, condom, or diaphragm) during the course of the trial. Oral birth control methods alone will not be considered adequate on this study, because of the potential pharmacokinetic interaction between study drug and oral contraceptives. Concomitant use of oral and barrier contraceptives is advised. Contraception is necessary for at least 6 months after receiving the study protein kinase inhibitor.
17. Concomitant medication with drugs having proarrhythmic potential (such as sotalol, haloperidol, flecainide) is not permitted during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12-27 (Actual); Study Completion 2017-12-27 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated plasma AUC0-12h of high-dose, pulsatile sorafenib | The exposure limiting toxicity period is within the first 42 days from the start of treatment. The maximum tolerated AUC0-12h of sorafenib is determined after completion of the escalation part of the study. It is expected to be completed within one year.
  Toxicity is graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events version 4.0.

SECONDARY OUTCOMES:
AUC0-12h of sorafenib and its primary active metabolite pyridine-N-oxide (escalation cohorts) | Pharmacokinetics analysis is performed during the first three treatment cycles (i.e. day 1, 8 en 15).
Cmax of sorafenib and its primary active metabolite pyridine-N-oxide (escalation cohorts) | Pharmacokinetics analysis is performed during the first three treatment cycles (i.e. day 1, 8 en 15).
Tmax of sorafenib and its primary active metabolite pyridine-N-oxide (escalation cohorts) | Pharmacokinetics analysis is performed during the first three treatment cycles (i.e. day 1, 8 en 15).
T1/2 of sorafenib and its primary active metabolite pyridine-N-oxide (escalation cohorts) | Pharmacokinetics analysis is performed during the first three treatment cycles (i.e. day 1, 8 en 15).
Recommended phase II dose | This depends on the maximum tolerated AUC0-12h of sorafenib. The maximum tolerated AUC0-12h of sorafenib is determined after completion of the escalation part of the study. It is expected to be completed within one year.
Preliminary efficacy i.e. response rate, progression free survival and overall survival. | From start of treatment until the date of death from any cause, assessed up to 100 months
  In an expansion cohort, 10 extra patients will be treated with high-dose, pulsatile sorafenib administrated at the maximum tolerated AUC. Before treatment and every 8 weeks during treatment CT thorax and abdomen will be performed and evaluated according to RECIST version 1.1.
Intratumoral and skin concentrations of sorafenib | After 2 weeks of treatment.
  Biopsies are only mandatory in the patients included in the expansion cohort. Concentrations are measured in biopsies using LC/MS/MS.
Optimal timepoints for finger puncture to determine sorafenib exposure | The finger punctures will be performed during the first three cycles (i.e. at day 1, 8 and 15)
  Finger punctures are only mandatory in de patients included in the expansion cohort. The results of the finger puncture will be compared with plasma and whole blood venous PK samples used for the AUC0-12h. The aim is to simplify full pharmacokinetic AUC sampling and to develop a method that can easily guide dose-adjustments based on sorafenib exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Henk MW Verheul, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Strumberg D, Richly H, Hilger RA, Schleucher N, Korfee S, Tewes M, Faghih M, Brendel E, Voliotis D, Haase CG, Schwartz B, Awada A, Voigtmann R, Scheulen ME, Seeber S. Phase I clinical and pharmacokinetic study of the Novel Raf kinase and vascular endothelial growth factor receptor inhibitor BAY 43-9006 in patients with advanced refractory solid tumors. J Clin Oncol. 2005 Feb 10;23(5):965-72. doi: 10.1200/JCO.2005.06.124. Epub 2004 Dec 21. PMID 15613696
- [Background] Pecuchet N, Lebbe C, Mir O, Billemont B, Blanchet B, Franck N, Viguier M, Coriat R, Tod M, Avril MF, Goldwasser F. Sorafenib in advanced melanoma: a critical role for pharmacokinetics? Br J Cancer. 2012 Jul 24;107(3):455-61. doi: 10.1038/bjc.2012.287. Epub 2012 Jul 5. PMID 22767146
- [Background] Wang X, Zhang L, Goldberg SN, Bhasin M, Brown V, Alsop DC, Signoretti S, Mier JW, Atkins MB, Bhatt RS. High dose intermittent sorafenib shows improved efficacy over conventional continuous dose in renal cell carcinoma. J Transl Med. 2011 Dec 21;9:220. doi: 10.1186/1479-5876-9-220. PMID 22188900
- [Background] Honeywell R, Yarzadah K, Giovannetti E, Losekoot N, Smit EF, Walraven M, Lind JS, Tibaldi C, Verheul HM, Peters GJ. Simple and selective method for the determination of various tyrosine kinase inhibitors used in the clinical setting by liquid chromatography tandem mass spectrometry. J Chromatogr B Analyt Technol Biomed Life Sci. 2010 May 1;878(15-16):1059-68. doi: 10.1016/j.jchromb.2010.03.010. Epub 2010 Mar 15. PMID 20382575